CLINICAL TRIAL: NCT00430118
Title: ALL-BFM 2000 Multi-Center Study for the Treatment of Children and Adolescents With Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy Based on Risk of Relapse in Treating Young Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Martin Schrappe, Prof. Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000528029; ALL-BFM-2000; EU-20682
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Leukemia
Keywords: T-cell childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine; Vindesine; Radiotherapy

ARMS (10):
- Induction Prot I/Dexa - reinduction Prot III (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Pred - reinduction Prot III (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Dexa - reinduction Prot II (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Pred - reinduction Prot II (Active Comparator)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Dexa - reinduction 2x Prot III (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Pred - reinduction 2x Prot III (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Dexa - reinduction 3 HR courses + 3x Prot III (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Pred - reinduction 3 HR courses + 3x Prot III (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Dexa - reinduction 6 HR courses + Prot II (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy
- Induction Prot I/Pred - reinduction 6 HR courses + Prot II (Active Comparator)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Drug: vindesine; Radiation: radiation therapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide
  Arms: Induction Prot I/Dexa - reinduction 3 HR courses + 3x Prot III; Induction Prot I/Dexa - reinduction 6 HR courses + Prot II; Induction Prot I/Pred - reinduction 3 HR courses + 3x Prot III; Induction Prot I/Pred - reinduction 6 HR courses + Prot II
Drug: ifosfamide
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisone
Drug: thioguanine
Drug: vincristine sulfate
Drug: vindesine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating young patients with acute lymphoblastic leukemia.

PURPOSE: Thisphase III trial is studying several different combination chemotherapy regimens to compare how well they work in treating young patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the relative efficacy of induction therapy comprising dexamethasone or prednisone, in terms of a higher rate of event-free survival (EFS) and overall survival and a reduced rate of relapse, in pediatric patients with intermediate-risk or high-risk acute lymphoblastic leukemia (ALL).
* Compare the relative safety of a reduced-intensity reintensification regimen comprising dexamethasone, vincristine, cyclophosphamide, and anthracyclines vs a standard treatment regimen in pediatric patients with standard-risk ALL identified by fast clearance of leukemic cells.
* Compare the efficacy of a second delayed reintensification regimen vs standard reintensification therapy, in terms of improved EFS, in pediatric patients with intermediate-risk ALL.
* Compare the efficacy of extended reintensification therapy (triple reinduction) vs standard reintensification therapy (intensive pulses and one reintensification) in pediatric patients with high-risk ALL.

OUTLINE: This is a randomized, multicenter study.

* Prednisone prephase therapy: Patients receive oral prednisone on days 1-7 and one dose of methotrexate (MTX) intrathecally (IT) on day 1.
* Induction/consolidation therapy, protocol I: Patients are randomized to 1 of 2 treatment arms.

  * Arm I (closed to accrual as of 6/30/2006): Patients receive prednisone (PRED) on days 8-28.
  * Arm II (closed to accrual as of 6/30/2006): Patients receive dexamethasone (DEXA) on days 8-28.

Patients in both arms also receive vincristine (VCR) and daunorubicin hydrochloride (DNR) once weekly in weeks 2-5; asparaginase (ASP) on days 12-33; cyclophosphamide (CPM) on days 36 and 64; cytarabine (ARA-C) in weeks 6-9; mercaptopurine (MP) on days 36-63; and MTX IT on days 1, 12, 33, 45, and 59.*

NOTE: *Patients with CNS disease also receive MTX IT on days 18 and 27.

After completion of induction/consolidation therapy, patients are stratified according to risk group based on disease response (standard-risk [SR] group [negative minimal residual disease (MRD) on day 33 and before protocol M, day 78] vs high-risk [HR] group [MRD ≥ 10^-³ on day 78] vs intermediate-risk [IR] group [all nonSR/nonHR]).* Patients with SR and IR disease proceed to extracompartment therapy. Patients with HR disease proceed to reintensification therapy.

NOTE: *Patients meeting any of the following criteria are placed in the HR group regardless of MRD response: Philadelphia chromosome-positive disease (BCR/ABL or t[9;22]; translocations [t4;11][q11;q23] or MLL/AF4); "prednisone-poor-response" (≥ 1,000 blasts/mm³ in the peripheral blood on day 8 after prednisone prephase therapy); or no response to study induction therapy (M2/3 at day 33).

* Extracompartment therapy, protocol M: Patients receive MP on days 1-56 and MTX on days 8, 22, 36, and 50.

After completion of extracompartment therapy, SR and IR patients proceed to reintensification therapy. SR patients are randomized to arms I or II. IR patients are randomized to arms I or III. HR patients who have completed induction/consolidation therapy are randomized to arms IV or V.

* Reintensification therapy:

  * Arm I (standard reinduction therapy, protocol II [closed to accrual as of 6/30/2006]): SR and IR patients receive DEXA on days 1-22; VCR and doxorubicin hydrochloride (DOX) in weeks 2-5; ASP on days 8, 11, 15, and 18; CPM on day 36; ARA-C and thioguanine (TG) on days 36-49; and MTX IT on days 38 and 45.* Patients then proceed to maintenance therapy.

NOTE: *Patients with CNS disease also receive MTX IT on days 1 and 18.

* Arm II (reduced-intensity reinduction therapy, protocol III [closed to accrual as of 6/30/2006]): SR patients receive DEXA on days 1-15; VCR and DOX on days 1 and 8; ASP on days 1, 4, 8, and 11; CPM on day 15; ARA-C and TG on days 15-28; and MTX IT on days 17 and 24.* Patients then proceed to maintenance therapy.

NOTE: *Patients with CNS disease also receive MTX on day 1.

* Arm III (reduced-intensity reinduction/second delayed reinduction therapy [double reintensification therapy] [closed to accrual as of 6/30/2006]): IR patients receive reduced-intensity reintensification therapy as in arm II. After a 10-week interim maintenance phase, treatment repeats once for a second delayed course of reintensification therapy. Patients then proceed to maintenance therapy.
* Arm IV (standard reintensification therapy [closed to accrual as of 6/30/2006]): HR patients receive two sequences of the following HR therapy elements (i.e., in this order: 1, 2, 3, 1, 2, 3) following reintensification therapy as in arm I. Patients then proceed to maintenance therapy.

  * Element HR-1: Patients receive DEXA on days 1-5; VCR on days 1 and 6; ARA-C twice on day 5; MTX and CPM every 12 hours on days 2-4 (5 doses); ASP on days 6 and 11; and MTX/ARA-C/PRED IT on day 1.
  * Element HR-2: Patients receive DEXA on days 1-5; vindesine on days 1 and 6; DNR on day 5; MTX and ifosfamide every 12 hours on days 2-4 (5 doses); ASP on days 6 and 11; and MTX/ARA-C/PRED IT on day 1.* NOTE: *HR patients with CNS disease also receive IT therapy on day 5.
  * Element HR-3: Patients receive DEXA on days 1-5; ARA-C every 12 hours on days 1-2 (4 doses); etoposide five times daily on days 3-5; ASP on days 6 and 11; and MTX/ARA-C/PRED IT on day 1.
* Arm V (extended reintensification therapy [triple protocol III] [closed to accrual as of 6/30/2006]): HR patients receive HR therapy elements 3, 2, and 1 as in arm IV following reintensification therapy as in arm II repeated the therapy element twice with 4-week interim maintenance phases in between. Patients then proceed to maintenance therapy.

  * Interim maintenance/maintenance therapy: Patients receive MTX once weekly and MP daily until week 104.
  * Radiotherapy: HR patients or patients with T-cell acute lymphoblastic leukemia or CNS disease undergo CNS radiotherapy.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute lymphoblastic leukemia (ALL)
* No secondary ALL

PATIENT CHARACTERISTICS:

* No prior disease that would preclude treatment with chemotherapy

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy
* More than 4 weeks since prior steroids

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4559 (Actual)
Dates: Start 2000-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of dexamethasone vs prednisone during the induction phase | End of Trial
Event-free survival (EFS) and overall survival after initial remission in intermediate-risk and high-risk patients | End of Trial
Safety and efficacy of treatment reduction during reintensification in standard-risk patients | End of Trial
EFS after second delayed reintensification in intermediate-risk patients | End of Trial
Outcome after extended reintensification therapy in high-risk patients | End of Trial

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schrappe, MD, PhD, Study Chair — University Hospital Schleswig-Holstein
Locations (76):
- Austria (10):
  - Krankenhaus Dornbirn, Dornbirn
  - Landeskrankenhaus Feldkirch, Feldkirch-Tisis
  - Universitaet Kinderklinik, Graz
  - Innsbruck Universitaetsklinik, Innsbruck
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - LKH Leoben, Leoben
  - A. oe. Krankenhaus der Barmherzigen Schwestern Kinderabteilung, Linz
  - Landes-Kinderkrankenhaus, Linz
  - St. Johanns-Spital, Salzburg
  - St. Anna Children's Hospital, Vienna
- Germany (60):
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Caritas-Krankenhaus Bad Mergentheim, Bad Mergentheim
  - Klinikum Bayreuth, Bayreuth
  - Helios Klinikum Berlin, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Kinderklinik der Universitaet Bonn, Bonn
  - Staedtisches Klinikum - Howedestrase, Braunschweig
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Coburg, Coburg
  - Kliniken der Stadt Koeln gGmbH - Kinderkrankenhaus Riehl, Cologne
  - Children's Hospital, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Vestische Kinderklinik Universitaetsklinik Witten/Herdecke, Datteln
  - Klinikum Lippe - Detmold, Detmold
  - Klinikum Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Klinikum Duisburg, Duisburg
  - Helios Klinikum Erfurt, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Kinderklinik, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitaetsklinikum Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - SLK - Kliniken Heilbronn GmbH - Klinikum am Gesundbrunnen, Heilbronn
  - Gemeinschaftskrankenhaus, Herdecke
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaets - Kinderklinik, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinikum Kemperhof Koblenz, Koblenz
  - St. Annastift Krankenhaus, Ludwigshafen
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitatsklinikum der MA, Magdeburg
  - Staedtisches Klinik - Kinderklinik, Mannheim
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Klinikum Minden, Minden
  - Krankenhaus Muenchen Schwabing, Munich
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Kinderklinik Kohlhof, Neunkirchen
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Kinderklinik - Universitaetsklinikum Rostock, Rostock
  - Saarbrucker Winterbergkliniken, Saarbrücken
  - Johanniter-Kinderklinik, Sankt Augustin
  - Klinikum Schwerin, Schwerin
  - Kinderklink Siegen Deutsches Rotes Kreuz, Siegen
  - Olgahospital, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Reinhard-Nieter-Krankenhaus, Wilhelmshaven
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Switzerland (6):
  - Kantonsspital Aarau, Aarau
  - Universitaets-Kinderspital beider Basel, Basel
  - Ospedale "la Carita", Locarno, Locarno
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital, Zurich

REFERENCES:
- [Background] Attarbaschi A, Mann G, Panzer-Grumayer R, Rottgers S, Steiner M, Konig M, Csinady E, Dworzak MN, Seidel M, Janousek D, Moricke A, Reichelt C, Harbott J, Schrappe M, Gadner H, Haas OA. Minimal residual disease values discriminate between low and high relapse risk in children with B-cell precursor acute lymphoblastic leukemia and an intrachromosomal amplification of chromosome 21: the Austrian and German acute lymphoblastic leukemia Berlin-Frankfurt-Munster (ALL-BFM) trials. J Clin Oncol. 2008 Jun 20;26(18):3046-50. doi: 10.1200/JCO.2008.16.1117. PMID 18565891
- [Result] Schrappe M, Valsecchi MG, Bartram CR, Schrauder A, Panzer-Grumayer R, Moricke A, Parasole R, Zimmermann M, Dworzak M, Buldini B, Reiter A, Basso G, Klingebiel T, Messina C, Ratei R, Cazzaniga G, Koehler R, Locatelli F, Schafer BW, Arico M, Welte K, van Dongen JJ, Gadner H, Biondi A, Conter V. Late MRD response determines relapse risk overall and in subsets of childhood T-cell ALL: results of the AIEOP-BFM-ALL 2000 study. Blood. 2011 Aug 25;118(8):2077-84. doi: 10.1182/blood-2011-03-338707. Epub 2011 Jun 30. PMID 21719599
- [Result] Conter V, Bartram CR, Valsecchi MG, Schrauder A, Panzer-Grumayer R, Moricke A, Arico M, Zimmermann M, Mann G, De Rossi G, Stanulla M, Locatelli F, Basso G, Niggli F, Barisone E, Henze G, Ludwig WD, Haas OA, Cazzaniga G, Koehler R, Silvestri D, Bradtke J, Parasole R, Beier R, van Dongen JJ, Biondi A, Schrappe M. Molecular response to treatment redefines all prognostic factors in children and adolescents with B-cell precursor acute lymphoblastic leukemia: results in 3184 patients of the AIEOP-BFM ALL 2000 study. Blood. 2010 Apr 22;115(16):3206-14. doi: 10.1182/blood-2009-10-248146. Epub 2010 Feb 12. PMID 20154213
- [Result] Kox C, Zimmermann M, Stanulla M, Leible S, Schrappe M, Ludwig WD, Koehler R, Tolle G, Bandapalli OR, Breit S, Muckenthaler MU, Kulozik AE. The favorable effect of activating NOTCH1 receptor mutations on long-term outcome in T-ALL patients treated on the ALL-BFM 2000 protocol can be separated from FBXW7 loss of function. Leukemia. 2010 Dec;24(12):2005-13. doi: 10.1038/leu.2010.203. Epub 2010 Oct 14. PMID 20944675
- [Result] Schrey D, Borghorst S, Lanvers-Kaminsky C, Hempel G, Gerss J, Moricke A, Schrappe M, Boos J. Therapeutic drug monitoring of asparaginase in the ALL-BFM 2000 protocol between 2000 and 2007. Pediatr Blood Cancer. 2010 Jul 1;54(7):952-8. doi: 10.1002/pbc.22417. PMID 20108339
- [Result] Dworzak MN, Schumich A, Printz D, Potschger U, Husak Z, Attarbaschi A, Basso G, Gaipa G, Ratei R, Mann G, Gadner H. CD20 up-regulation in pediatric B-cell precursor acute lymphoblastic leukemia during induction treatment: setting the stage for anti-CD20 directed immunotherapy. Blood. 2008 Nov 15;112(10):3982-8. doi: 10.1182/blood-2008-06-164129. Epub 2008 Sep 9. PMID 18780832
- [Result] Flohr T, Schrauder A, Cazzaniga G, Panzer-Grumayer R, van der Velden V, Fischer S, Stanulla M, Basso G, Niggli FK, Schafer BW, Sutton R, Koehler R, Zimmermann M, Valsecchi MG, Gadner H, Masera G, Schrappe M, van Dongen JJ, Biondi A, Bartram CR; International BFM Study Group (I-BFM-SG). Minimal residual disease-directed risk stratification using real-time quantitative PCR analysis of immunoglobulin and T-cell receptor gene rearrangements in the international multicenter trial AIEOP-BFM ALL 2000 for childhood acute lymphoblastic leukemia. Leukemia. 2008 Apr;22(4):771-82. doi: 10.1038/leu.2008.5. Epub 2008 Jan 31. PMID 18239620
- [Derived] Junk SV, Schaeffeler E, Zimmermann M, Moricke A, Beier R, Schutte P, Fedders B, Alten J, Hinze L, Klein N, Kulozik A, Muckenthaler MU, Koehler R, Borkhardt A, Vijayakrishnan J, Ellinghaus D, Forster M, Franke A, Wintering A, Kratz CP, Schrappe M, Schwab M, Houlston RS, Cario G, Stanulla M. Chemotherapy-related hyperbilirubinemia in pediatric acute lymphoblastic leukemia: a genome-wide association study from the AIEOP-BFM ALL study group. J Exp Clin Cancer Res. 2023 Jan 13;42(1):21. doi: 10.1186/s13046-022-02585-x. PMID 36639636
- [Derived] Stanulla M, Dagdan E, Zaliova M, Moricke A, Palmi C, Cazzaniga G, Eckert C, Te Kronnie G, Bourquin JP, Bornhauser B, Koehler R, Bartram CR, Ludwig WD, Bleckmann K, Groeneveld-Krentz S, Schewe D, Junk SV, Hinze L, Klein N, Kratz CP, Biondi A, Borkhardt A, Kulozik A, Muckenthaler MU, Basso G, Valsecchi MG, Izraeli S, Petersen BS, Franke A, Dorge P, Steinemann D, Haas OA, Panzer-Grumayer R, Cave H, Houlston RS, Cario G, Schrappe M, Zimmermann M; TRANSCALL Consortium; International BFM Study Group. IKZF1plus Defines a New Minimal Residual Disease-Dependent Very-Poor Prognostic Profile in Pediatric B-Cell Precursor Acute Lymphoblastic Leukemia. J Clin Oncol. 2018 Apr 20;36(12):1240-1249. doi: 10.1200/JCO.2017.74.3617. Epub 2018 Mar 2. PMID 29498923
- [Derived] Schrappe M, Bleckmann K, Zimmermann M, Biondi A, Moricke A, Locatelli F, Cario G, Rizzari C, Attarbaschi A, Valsecchi MG, Bartram CR, Barisone E, Niggli F, Niemeyer C, Testi AM, Mann G, Ziino O, Schafer B, Panzer-Grumayer R, Beier R, Parasole R, Gohring G, Ludwig WD, Casale F, Schlegel PG, Basso G, Conter V. Reduced-Intensity Delayed Intensification in Standard-Risk Pediatric Acute Lymphoblastic Leukemia Defined by Undetectable Minimal Residual Disease: Results of an International Randomized Trial (AIEOP-BFM ALL 2000). J Clin Oncol. 2018 Jan 20;36(3):244-253. doi: 10.1200/JCO.2017.74.4946. Epub 2017 Nov 17. PMID 29148893
- [Derived] Zuna J, Moericke A, Arens M, Koehler R, Panzer-Grumayer R, Bartram CR, Fischer S, Fronkova E, Zaliova M, Schrauder A, Stanulla M, Zimmermann M, Trka J, Stary J, Attarbaschi A, Mann G, Schrappe M, Cario G. Implications of delayed bone marrow aspirations at the end of treatment induction for risk stratification and outcome in children with acute lymphoblastic leukaemia. Br J Haematol. 2016 Jun;173(5):742-8. doi: 10.1111/bjh.13989. Epub 2016 Feb 23. PMID 26913693
- [Derived] Moricke A, Zimmermann M, Valsecchi MG, Stanulla M, Biondi A, Mann G, Locatelli F, Cazzaniga G, Niggli F, Arico M, Bartram CR, Attarbaschi A, Silvestri D, Beier R, Basso G, Ratei R, Kulozik AE, Lo Nigro L, Kremens B, Greiner J, Parasole R, Harbott J, Caruso R, von Stackelberg A, Barisone E, Rossig C, Conter V, Schrappe M. Dexamethasone vs prednisone in induction treatment of pediatric ALL: results of the randomized trial AIEOP-BFM ALL 2000. Blood. 2016 Apr 28;127(17):2101-12. doi: 10.1182/blood-2015-09-670729. Epub 2016 Feb 17. PMID 26888258
- [Derived] Cario G, Rhein P, Mitlohner R, Zimmermann M, Bandapalli OR, Romey R, Moericke A, Ludwig WD, Ratei R, Muckenthaler MU, Kulozik AE, Schrappe M, Stanulla M, Karawajew L. High CD45 surface expression determines relapse risk in children with precursor B-cell and T-cell acute lymphoblastic leukemia treated according to the ALL-BFM 2000 protocol. Haematologica. 2014 Jan;99(1):103-10. doi: 10.3324/haematol.2013.090225. Epub 2013 Aug 2. PMID 23911702
- [Derived] Dorge P, Meissner B, Zimmermann M, Moricke A, Schrauder A, Bouquin JP, Schewe D, Harbott J, Teigler-Schlegel A, Ratei R, Ludwig WD, Koehler R, Bartram CR, Schrappe M, Stanulla M, Cario G. IKZF1 deletion is an independent predictor of outcome in pediatric acute lymphoblastic leukemia treated according to the ALL-BFM 2000 protocol. Haematologica. 2013 Mar;98(3):428-32. doi: 10.3324/haematol.2011.056135. Epub 2012 Aug 8. PMID 22875627
- [Derived] Zeidler L, Zimmermann M, Moricke A, Meissner B, Bartels D, Tschan C, Schrauder A, Cario G, Goudeva L, Jager S, Ratei R, Ludwig WD, Teigler-Schlegel A, Skokowa J, Koehler R, Bartram CR, Riehm H, Schrappe M, Welte K, Stanulla M. Low platelet counts after induction therapy for childhood acute lymphoblastic leukemia are strongly associated with poor early response to treatment as measured by minimal residual disease and are prognostic for treatment outcome. Haematologica. 2012 Mar;97(3):402-9. doi: 10.3324/haematol.2011.045229. Epub 2011 Nov 4. PMID 22058224
- [Derived] Willer A, Gerss J, Konig T, Franke D, Kuhnel HJ, Henze G, von Stackelberg A, Moricke A, Schrappe M, Boos J, Lanvers-Kaminsky C. Anti-Escherichia coli asparaginase antibody levels determine the activity of second-line treatment with pegylated E coli asparaginase: a retrospective analysis within the ALL-BFM trials. Blood. 2011 Nov 24;118(22):5774-82. doi: 10.1182/blood-2011-07-367904. Epub 2011 Sep 22. PMID 21940824